CLINICAL TRIAL: NCT06206421
Title: A Phase 3, Randomized, Placebo-controlled, Double-blind Study to Investigate the Long Term Safety of Fezolinetant in Japanese Women Suffering From Vasomotor Symptoms (Hot Flashes) Associated With Menopause
Brief Title: A Study to Assess Long-term Safety of Fezolinetant Given to Japanese Women Going Through Menopause
Acronym: Starlight 3
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2693-CL-0311; jRCT2031230584 (Registry Identifier: jRCT)
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Hot Flashes
Keywords: menopause;; ESN364;; vasomotor symptoms;; fezolinetant;; VEOZAH™
MeSH Terms: conditions — Hot Flashes | interventions — fezolinetant

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fezolinetant (Experimental): Participants will receive fezolinetant once daily for 52 weeks.
  Interventions: Drug: Fezolinetant
- Placebo (Experimental): Participants will receive matching placebo once daily for 52 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fezolinetant — oral
  Other Names: ESN364;; VEOZAH™
  Arms: Fezolinetant
Drug: Placebo — oral
  Arms: Placebo

SUMMARY:
Hot flashes are the most common reason women going through menopause seek medical attention. Hormone replacement therapy, or HRT, is most often prescribed to treat hot flashes. However, HRT can't be used by all women or for as long as may be needed.

Researchers want to find other ways to treat hot flashes. Fezolinetant is a medicine to treat hot flashes in women going through menopause. Fezolinetant is an approved medicine in the US. Further studies are needed before it is available in other regions such as Asia.

In this study fezolinetant will be used to treat hot flashes in Japanese women going through menopause. This study will confirm the safety of fezolinetant and how well the women tolerate the treatment.

Women will either take fezolinetant or a placebo. This is decided by chance alone. The placebo looks like fezolinetant but will not have any medicine in it.

The women will take 1 tablet of the study medicine (fezolinetant or the placebo) once a day for up to 52 weeks.

During the study, the women will visit their study clinic for a check-up about every 4 weeks for up to 52 weeks (1 year). At each visit they will be asked if they had any medical problems. Other checks will include a medical examination and vital signs (temperature, blood pressure and pulse). At some visits, the women will have an ECG to check their heart rhythm and some blood and urine samples will be taken for laboratory tests. During a couple of visits, women who have a womb (uterus) will also have a test called a transvaginal ultrasound. A probe is gently placed inside the vagina. Sound waves will create a picture of the organs in the pelvis. This will allow the study doctor to look more closely at the uterus and surrounding organs.

The last clinic visit will be 3 weeks after the women take their final tablet of the study medicine (fezolinetant or the placebo).

ELIGIBILITY:
Inclusion Criteria:

* Participant confirmed as menopausal per one of the following criteria at the screening visit (visit 1):

  * For a post-menopausal participant: Spontaneous amenorrhea for >/=12 consecutive months; Spontaneous amenorrhea for >/=6 months with biochemical criteria of menopause (follicle-stimulating hormone (FSH) > 40 IU/L); Having had bilateral oophorectomy >/=6 weeks prior to the screening visit (visit 1) (with or without hysterectomy); Having had hysterectomy without bilateral oophorectomy with the biochemical criteria of menopause (FSH > 40 IU/L); or Having been confirmed to be post-menopausal in the 2693-CL-0310 study.
  * For a peri-menopausal participant: Spontaneous amenorrhea for >/=60 days but < 6 consecutive months 2 times in the 2 most recent menstrual cycles with biochemical criteria of peri-menopause (FSH > 25 IU/L); or Spontaneous amenorrhea for >/=6 months but < 12 consecutive months with biochemical criteria of peri-menopause (FSH > 25 IU/L and ≤ 40 IU/L); Having had hysterectomy without bilateral oophorectomy with the biochemical criteria of peri-menopause (FSH > 25 IU/L and ≤ 40 IU/L).
* Participant is seeking treatment for relief of vasomotor symptoms (VMS) associated with menopause.
* Female participant:

  * Is not pregnant and at least 1 of the following conditions apply: Not a women of childbearing potential (WOCBP); WOCBP who has a negative urine pregnancy test day 1 (visit 2) and agrees to follow the contraceptive guidance from the time of informed consent through at least 21 days after final study intervention administration.
  * Must not be breastfeeding or lactating starting at screening and throughout the investigational period and for 21 days after final study intervention administration.
  * Must not donate ova starting at first administration of study intervention and throughout the investigational period and for 21 days after final study intervention administration
* Participant agrees not to participate in another interventional study while participating in the present study.

Exclusion Criteria:

* Participant has a history of an undiagnosed uterine bleeding within the 6 months prior to the screening visit (visit 1).
* Participant has a current malignant tumor or history (except for a participant who has not received treatment for malignant tumors for at least 5 years before informed consent acquisition and was not considered to have recurrence) of a malignant tumor except for non-metastatic basal cell carcinoma of the skin.
* Participant has a medical condition or chronic disease (including history of neurological [including cognitive], hepatic, renal, cardiovascular, gastrointestinal, pulmonary [e.g., moderate asthma], endocrine, or gynecological disease) that could confound interpretation of the study outcome.
* Participant uses a prohibited therapy (hormone therapy, hormone replacement therapy (HRT), hormonal contraceptive, any treatment for VMS [prescription medications, over-the-counter, or herbal/Kampo medicines] or strong or moderate cytochrome P450 1A2 (CYP1A2) inhibitors and is not willing to wash out or discontinue use of such drugs from screening visit (visit 1) through the follow-up visit (visit 16) or it is not medically appropriate to discontinue such drugs for the duration of the study.
* Participant has been randomized/registered in a clinical trial with fezolinetant previously or had previous exposure to marketed fezolinetant elsewhere.
* Participant has a present or previous history of participation in this study.
* Participant has received any investigational therapy within 28 days or 5 half-lives, whichever is longer, prior to screening visit (visit 1).
* Participant has an unacceptable result from the transvaginal ultrasound (TVU) assessment at screening (i.e., full length of endometrial cavity cannot be visualized or presence of clinically significant abnormal findings).
* Participant has documentation of a clinically significant abnormal Papanicolaou (Pap) test (or equivalent cervical cytology) within 12 months prior to the screening visit (visit 1) or at screening.
* Participant has active liver disease, jaundice, or elevated liver aminotransferases (alanine aminotransferase (ALT) or aspartate aminotransferase (AST)), elevated total bilirubin (TBL) or direct bilirubin (DBL), elevated international normalized ratio (INR), or elevated alkaline phosphatase (ALP) at screening. A participant with mildly elevated ALT or AST up to < 1.5 × upper limit of normal (ULN) can be enrolled if TBL and DBL are normal. Participant with mildly elevated ALP (up to < 1.5 × ULN) can be enrolled if cholestatic liver disease is excluded and no cause other than fatty liver is diagnosed. Participant with Gilbert's syndrome with elevated TBL may be enrolled as long as DBL, hemoglobin and reticulocytes are normal.
* Participant has creatinine > 1.5 × ULN or estimated glomerular filtration rate using the Modification of Diet in Renal Disease formula </=30 mL/min/1.73 m^2 at screening.
* Participant has positive hepatitis serology panel (i.e., positive hepatitis B surface (HBs) antigen and/or positive hepatitis C virus (HCV) antibody) at screening. If HCV antibody test result is equivocal, hepatitis C virus ribonucleic acid (HCV RNA) test at study site is allowed. Participant can be enrolled if that result is normal or not abnormal.
* Participant is not in good general health as determined on the basis of medical history and general physical examination performed at the screening; hematology parameters, biochemistry parameters, pulse rate, blood pressure, electrocardiogram (ECG) outside the reference range for the population studied, or is showing clinically relevant deviations.
* Participant has a history of suicide attempt or suicidal behavior within 12 months prior to study enrollment or suicidal ideation within 12 months prior to study enrollment (a response of "yes" to question 4 or 5 on the suicidal ideation portion of the Columbia Suicide Severity Rating Scale (C-SSRS)), or is at significant risk to commit suicide at day 1 (visit 2).
* Participant is unable or unwilling to complete the study procedures.
* Participant has any condition which makes the participant unsuitable for study participation.
* Participant has a known or suspected hypersensitivity to fezolinetant or any components of the formulation used.
* Participant is the investigator or a member of the study site staff.
* Participant is an employee of Astellas, the study-related contract research organizations (CROs) or site management organizations.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2024-02-22 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) | Up to Week 55
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
  An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention. This includes events related to the comparator, if applicable, and events related to the (study) procedures.

SECONDARY OUTCOMES:
Change from baseline in endometrial thickness in post-menopausal participants | Baseline and up to Week 52
  Endometrial thickness is a measure of how thick the lining of the uterus is. Endometrial thickness will be measured by transvaginal ultrasound (TVU).
Number of participants with laboratory value abnormalities and/or AEs | Up to Week 55
  Number of participants with potentially clinically significant laboratory values.
Number of participants with vital sign abnormalities and/or AEs | Up to Week 55
  Number of participants with potentially clinically significant vital sign values.
Number of participants with electrocardiogram (ECG) abnormalities and/or AEs | Up to Week 52
  Number of participants with potentially clinically significant ECG values.
Pharmacokinetics (PK) of fezolinetant in plasma: Concentration | Up to Week 52
  Concentration will be recorded from the PK plasma samples collected.
Pharmacokinetics (PK) of metabolite ES259564 in plasma: Concentration | Up to Week 52
  Concentration will be recorded from the PK plasma samples collected.

CONTACTS AND LOCATIONS:
Overall Officials: Associate Medical Director, Study Director — Astellas Pharma Inc
Locations (24):
- Japan (24):
  - Daido Clinic, Nagoya, Aichi-ken
  - Juno Vesta Clinic hatta, Matsudo-shi, Chiba
  - Mori Ladies Clinic, Fukuoka, Fukuoka
  - Kotoni Ladies Clinic, Sapporo, Hokkaido
  - M's Ladies Clinic, Sapporo, Hokkaido
  - NISHIKAWA Women's Health Clinic, Sapporo, Hokkaido
  - Motomachi Ladies Clinic, Yokohama, Kanagawa
  - Women's Clinic LUNA Yokohama Motomachi, Yokohama, Kanagawa
  - Chieko Yukika Lady's Clinic, Sendai, Miyagi
  - GyNet Medical Corporation Minamimorimachi Ladies' Clinic, Osaka, Osaka
  - Ninomiya Ladies Clinic, Osaka, Osaka
  - Rikako Ladies Clinic, Osaka, Osaka
  - Tennoji Chihiro Women's Clinic, Osaka, Osaka
  - Shimizu Ladies Clinic, Sakai-shi, Osaka
  - jMOG Medical Corporation Tanabe Ladies' Clinic, Takatsuki-shi, Osaka
  - Marunouchi no Mori Ladies Clinic, Chiyoda-ku, Tokyo
  - Ginza Yoshida Medical Clinic, Chuo-ku, Tokyo
  - Medical Corporation Asbo Tokyo Asbo Clinic, Chuo-ku, Tokyo
  - Medical Corp.SEIKOUKAI New Medical Research System Clinic, Hachioji-shi, Tokyo
  - Kichijyoji Ladies Clinic, Musashino-shi, Tokyo
  - Shimamura Memorial Hospital, Nerima-ku, Tokyo
  - Yukawa Women'S Clinic, Nishi-Tokyo-shi, Tokyo
  - Shimodaira Ladies Clinic, Suginami-ku, Tokyo
  - Medical Corporation Associa Tamacenter Ladies Clinic, Tama-Shi, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/